CLINICAL TRIAL: NCT02905565
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Add-On to Standard Of-Care Study of n Butylphthalide (NBP) Softgel Capsules for Treatment of Mild to Moderate Acute Ischemic Stroke (AIS) in Adult Subjects
Brief Title: NBP in Adult Patients With Acute Ischemic Stroke (AIS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CSPC-NBP Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSPC-NBP-2001
Record Dates: First submitted 2016-08-23; First posted 2016-09-19 (Estimated); Last update posted 2020-09-17 (Actual); Status verified 2019-11

CONDITIONS: AIS
Keywords: Multicenter; Randomized; Double-Blind; Placebo-Controlled; Add-On to Standard-of-Care; Safety; Efficacy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Interventions: Placebo (NBP placebo softgel capsules, 0 mg NBP, BID)
  Interventions: Drug: Placebo
- 800 mg of NBP daily (Active Comparator): Interventions: 800 mg NBP softgel capsules daily (400 mg BID)
  Interventions: Drug: NBP Softgel Capsules

INTERVENTIONS:
Drug: NBP Softgel Capsules — Take 4 capsules BID on an empty stomach at least 1 hour before food intake, and remain fasting at least 1 hour after dosing.
  Other Names: NBP
  Arms: 800 mg of NBP daily
Drug: Placebo — Take 4 capsules BID on an empty stomach at least 1 hour before food intake, and remain fasting at least 1 hour after dosing
  Other Names: NBP Placebo Softgel Capsules
  Arms: Placebo

SUMMARY:
This is a Phase 2 multicenter, randomized, double-blind, placebo-controlled, add-on to standard of care study of NBP softgel capsules for the treatment of mild to moderate AIS in adults.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, add-on to standard-of-care study with a primary objective to assess the safety of NBP treatment in patients with mild to moderate acute ischemic stroke. The secondary objectives include determination of pharmacokinetic (PK) profile and exploratory evaluation for the efficacy of NBP treatment in stroke patients.

All randomized subjects will also receive standard supportive medical care for treatment of AIS throughout the study. The overall duration of the study will be approximately 90 days, including 30 days of treatment and an additional 60 days for follow up assessments. Subjects will be hospitalized long enough to receive the first four doses of study drug. After discharge from the hospital, subjects will continue to take study treatment daily through Day 30 and have scheduled assessments completed.

To maintain the blind, all subjects will take 4 softgel capsules BID, which will contain either 100 mg NBP or matching placebo. The first dose must be taken within 12 hours of the onset of the AIS defined as the last known normal.

ELIGIBILITY:
Inclusion Criteria

1. Males or females aged ≥ 18 and ≤ 85 years.
2. Women of childbearing potential (WOCBP) must have a negative urine human chorionic gonadotropin (HCG) pregnancy test at Screening and be practicing a medically acceptable method of contraception with an annual failure rate of less than 1% until the completion of the trial or 60 days after discontinuation of study treatment. Women are considered not childbearing if they are > 1 year postmenopausal or surgically sterile (ie, hysterectomy, bilateral oophorectomy, or bilateral salpingectomy tubal ligation). If serum beta human chorionic gonadotropin (bHCG) is the standard of care, then this value can be used to determine eligibility.
3. A clinical diagnosis of mild to moderate cortical or subcortical AIS.
4. Able to swallow the softgel capsules as defined by the investigator.
5. Completes screening procedures such that study treatment is first administered within 24 hours of stroke onset. The stroke onset time will be defined as the last known normal.
6. If Tissue Plasminogen Activator (tPA) is given as part of standard of care, the first dose of NBP must be administered no sooner than 4 hours after the end of the tPA infusion.
7. A standard NIHSS score of 4 to 17, inclusive. If patients receive tPA and/or endovascular treatment (EVT), the NIHSS score must be obtained after the infusion and/or procedure is completed. If sedation is used for EVT, then the NIHSS score must be obtained after sedation no longer confounds the assessment. All subjects must meet a NIHSS consciousness score of 0-1 in order to meet eligibility.
8. Functionally independent, as defined by a Modified Rankin Scale (mRS) score of 0 to 1 before their present illness as determined by the subject or provided by a representative if the subject is unable to participate at the time of study entry (determined by retrospective assessment by the Investigator).
9. Capable of understanding the purpose and risk of the study and has signed, in writing, the Informed Consent Form (ICF). If the subject is not capable of this at the time of enrollment, a legally authorized representative (LAR) will provide written informed consent in accordance with all regulations.
10. Ability to comply with study requirements.

Exclusion Criteria:

1. Female subjects who are pregnant, lactating/breast-feeding, or plan to become pregnant within the next 3 months.
2. Suspected diagnosis of stroke isolated to brainstem or brain areas other than cortical or subcortical AIS that may have caused the present symptoms, based on the opinion of the Investigator.
3. Rapidly improving or resolving symptoms, suggesting a possible transient ischemic attack (TIA) rather than a qualifying stroke.
4. Signs of acute intracranial hemorrhage or symptomatic hemorrhagic transformation of AIS defined by a 4-point worsening in NIHSS from presentation, or other cause of acute stroke symptoms (other than early ischemic findings) on cranial imaging at Screening.
5. History of intracranial hemorrhage.
6. Seizure at onset of stroke.
7. A previous clinical diagnosis of stroke within 6 months of current AIS. A previously undiagnosed stroke evidenced on screening CT or MRI may be enrolled provided it does not affect neurological and functional assessments based on the opinion of the Investigator.
8. Uncontrolled severe hypertension defined as a systolic blood pressure (SBP) ≥ 220 mm Hg or diastolic blood pressure (DBP) ≥ 110 mm Hg.
9. Treatment with intensive antihypertensive therapy within 4 hours of randomization.
10. SBP < 100 mm Hg, temperature > 38.0º C, or heart rate < 40 beats/minute or > 120 beats/minute at Screening or prior to randomization.
11. A glucose level of < 50 mg/dL at Screening.
12. An international normalized ratio (INR) ≥ 1.5 if not being treated with anticoagulant therapy, or an INR ≥ 3.5 if being treated with an acceptable anticoagulant therapy.
13. A serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level > 1.5 × Upper Limits of Normal (ULN), or bilirubin > 1.5 ULN (except in setting of known Gilbert's disease) at Screening.
14. Clinically significant renal dysfunction (including serum creatinine level > 2.0 mg/dL or 177 µmol/L) at Screening.
15. A hemoglobin level < 10 g/dL at Screening.
16. Current or within the last 6 months prior to Screening, New York Heart Association Class III/IV heart failure, severe uncorrected valve disease, known or suspected infective/vegetative endocarditis, ventricular tachycardia, or torsade de pointes.
17. Corrected QTcF (Fridericia) > 450 ms for male subjects or > 470 ms for female subjects (average of 3 ECG tracings) prior to randomization.
18. Current diagnosis of cancer or is being treated or has received any treatments for cancer within the last 5 years except basal cell carcinoma or curatively resected squamous cell carcinoma.
19. Known life expectancy < 6 months (for any reason).
20. Known allergy or hypersensitivity to celery or soybeans.
21. Received treatment with any other investigational drug within 30 days before Baseline, was previously treated with NBP, is currently taking celery seed extract, or is currently participating in another clinical study.
22. Known or suspected history of alcohol or drug dependence within the past 6 months, or is known to have abused alcohol (eg, been intoxicated) within the last 24 hours.
23. Known history of hepatitis B, hepatitis C, HIV, or tuberculous (TB).
24. Any other reasons that, in the opinion of the investigator, make the subject unsuitable for enrollment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2020-08-07 (Actual); Study Completion 2020-08-07 (Actual)

PRIMARY OUTCOMES:
Incidence rate of treatment-emergent adverse events (TEAEs) | 90 days
  Safety will be evaluated through the collection of TEAEs, serious adverse events (SAEs), clinical laboratory assessments, vital sign measurements, 12-lead ECGs, and physical and neurologic examinations. Suicidality will be evaluated at each clinical visit using the Columbia-Suicide Severity Rating Scale (C-SSRS).

SECONDARY OUTCOMES:
PK profile of NBP treatment in subjects with AIS | 1 day
  Peak and trough levels of NBP and metabolites
Exploratory efficacy outcome: mRS | 90 days
  Improvement of disability as measured by the mRS at Day 30 and Day 90
Exploratory efficacy outcome: Barthel Index (BI) Assessment | 90 days
  Stroke recovery as measured by the BI Assessment at Day 30 and Day 90
Exploratory efficacy outcome: NIHSS | 90 days
  Stroke recovery as measured by the NIHSS at Day 30 and Day 90
Exploratory efficacy outcome: Stroke Impact Scale (SIS) Assessment | 90 days
  SIS-16 on study Day 30 and 90

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Clarke, MD, Principal Investigator — Oregon Health and Science University
Locations (18):
- United States (18):
  - Investigative Site, Los Angeles, California
  - Investigative Site, Jacksonville, Florida
  - Investigative Site, Des Moines, Iowa
  - Investigative Site, Louisville, Kentucky
  - Investigative Site, Boston, Massachusetts
  - Investigative Site, Golden Valley, Minnesota
  - Investigative Site, St Louis, Missouri
  - Investigative Site, Omaha, Nebraska
  - Investigative Site, Buffalo, New York
  - Investigative Site, Asheville, North Carolina
  - Investigative Site, Columbus, Ohio
  - Investigative Site, Hillsboro, Oregon
  - Investigative Site, Portland, Oregon
  - Investigative Site, Philadelphia, Pennsylvania
  - Investigative Site, Charleston, South Carolina
  - Investigative Site, Columbia, South Carolina
  - Investigative Site, Chattanooga, Tennessee
  - Investigative Site, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No